CLINICAL TRIAL: NCT07145762
Title: Validity of the Analgesia Nociception Index in Children and Adolescents With Chronic Pain
Brief Title: Analgesia Nociception Index In Pediatric Patients With Chronic Pain
Acronym: Chronic pain
Status: Not yet recruiting | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Sabrina Carrie, Pediatric Anesthetist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: ANI Project
Record Dates: First submitted 2025-08-18; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic pain patients receiving Interventional block
  Interventions: Procedure: Interventional Block

INTERVENTIONS:
Procedure: Interventional Block — For patients who are offered interventional blocks as part of their standard of care, we will measure ANI as well as pressure pain threshold before, during, and after the block as well and at follow-up to assess correlation with treatment efficacy.

SUMMARY:
The goal of this observational study is to learn about the analgesia nociceptive index (ANI) is associated with pain sensitivity in patients between the ages of 9-17 who are experiencing chronic pain. The main question it aims to answer is:

- Does the ANI score correlate with the change in the pain sensitivity in patients aged 9-17 undergoing an interventional block.

Patients already receiving an interventional block as part of their regular medical care for chronic pain will have their level of pain recorded during clinic appointments

ELIGIBILITY:
Inclusion Criteria:

* Experiencing chronic pain defined by: persistent or recurrent pain at least once a week for at least three months in their electronic medical charts or by reference of the patient's physician

Exclusion Criteria:

* Taking medications known to affect the sympathetic or parasympathetic nervous systems such as cholinomimetics (e.g., pilocarpine), anticholinergics (e.g., ipratropium), sympathomimetics (e.g., salbutamol), and adrenergic antagonists (e.g., propranolol).
* Diagnosed cardiac or neurological conditions, including patients with arrhythmias, heart block, postural orthostatic tachycardia syndrome, Guillain-Barre syndrome, or spinal cord injury.
* Active cancer diagnosis
* Conditions that may interfere with the ability to understand instructions or complete assessments including: cognitive, or developmental delay.
* Patients who do not speak English or French.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients who are offered an interventional block at the Edwards Family Interdisciplinary Center for Complex Pain of the Montreal Children's Hospital will be invited to participate. Initial contact will be through the medical team in contact with the patient. They will ask them if they agree to be contacted for a research study. Once the patient consents to be contacted, the research coordinators will reach out the patient and explain the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Validation of analgesia nociception index (ANI) as a tool to assess change in the pain pressure threshold (PTT), measured by the PPT test, of children with chronic pain conditions. | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No